CLINICAL TRIAL: NCT01543607
Title: Endoscopic Therapy of Malignant Bile Duct Strictures: A Pilot Study
Brief Title: Endoscopic Therapy of Malignant Bile Duct Strictures
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, William R. Brugge, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-405
Record Dates: First submitted 2012-02-15; First posted 2012-03-05 (Estimated); Results first posted 2017-04-24 (Actual); Last update posted 2017-04-24 (Actual); Status verified 2017-03

CONDITIONS: Obstruction of Biliary Tree; Biliary Tract Cancer; Biliary Tract Neoplasms
Keywords: Bile duct; Cholangiocarcinoma; Bile duct stenosis; Malignant bile duct obstruction; Malignant bile duct stricture; Radiofrequency ablation; RFA; Endoscopic RFA catheter; EndoHPB
MeSH Terms: conditions — Biliary Tract Neoplasms; Cholangiocarcinoma | interventions — Catheter Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental): Radiofrequency ablation catheter
  Interventions: Device: Radiofrequency ablation catheter (Habib EndoHBP)

INTERVENTIONS:
Device: Radiofrequency ablation catheter (Habib EndoHBP) — Catheter placement into bile duct
  Other Names: Habib EndoHBP

SUMMARY:
Patients with malignant bile duct stenosis have poor prognosis and most of the patients are not good candidate for surgery at the time of diagnosis. Placement of the stent is the palliative care for these patients. However over 50% of the stents get blocked within 6-8 months. Use of the radiofrequency ablation before the stent placement may improve stent patency. Heat will be applied to the bile duct in order to open the blockage and prevent the re-growth of tissue into the stent. The investigators are looking to see how safe and feasible RFA (Radiofrequency ablation) catheter is in patient with malignant bile duct stenosis.

DETAILED DESCRIPTION:
As part of medical care subjects will be undergoing an endoscopic procedure (ERCP) in order to evaluate and stent a bile duct blockage. During the ECRP and just prior to the stent placement subjects will undergo the placement of a radiofrequency ablation catheter into the bile duct blockage. Heat will be applied to the bile duct in order to open the blockage and prevent the re-growth of tissue into the stent; after the radiofrequency ablation, stent will be placed. Three days after the procedure subjects will receive a phone call from the research coordinator to check any adverse or unwanted effects of the treatment. The study procedure (radiofrequency ablation) takes place over 10 minutes during ERCP. The subjects will undergo routine follow up for their medical problems. No follow up visits are required as part of the study.

ELIGIBILITY:
Inclusion Criteria:

* Documented malignant biliary obstruction requiring ERCP guided stenting

Exclusion Criteria:

* Coagulopathy (INR > 2.0 or PTT > 100 sec or platelet count < 50,000)
* Evidence of high-grade symptomatic duodenal obstruction
* Poor performance status
* Active suppurative cholangitis
* Complex stenoses will not be eligible for the trial
* Patients without access to duodenum or ampulla are not candidates for ERCP and stenting
* Candidates for a Whipple resection
* Patients who do not speak English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2012-02 (Actual); Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William R Brugge, M.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- See also: Study information — http://crnet.mgh.harvard.edu/trials.aspx?tId=4702

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Safety: Number of Bile Leak After RFA Procedure
Description: Determination of safety will be measured by the presence of a bile leak( bile leak will be defined by contrast cholangiography)
Time Frame: 2 years
Measure: Number; unit: bile leak
Arm/Group | Treatment
Number analyzed (Participants) | 1
bile leak | 1

2. Secondary Outcome: Feasibility: Ease of the Radiofrequency Ablation Catheter Placement
Description: Determine the feasibility of radiofrequency ablation catheter placement across malignant strictures with using a subjective scale, 0 is being impossible to place the catheter and 10 is being very easy to place the catheter.
Time Frame: 2 years
Measure: Number; unit: units on a scale
Arm/Group | Treatment
Number analyzed (Participants) | 1
units on a scale | 10

3. Secondary Outcome: Effectiveness: Change From Baseline in Bile Duct Diameter.
Description: Effectiveness will be determined by change in stricture diameter (increase or decrease) after RFA procedure. This will be measure as percentage change in improvement of the stricture.
Time Frame: 2 years
Measure: Number; unit: percentage of improvement:
Arm/Group | Treatment
Number analyzed (Participants) | 1
percentage of improvement: | 50

ADVERSE EVENTS:
Time Frame: 2 years.
Arm/Group | Treatment
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes